CLINICAL TRIAL: NCT04986748
Title: Q-SAM (Using QPOP to Predict Treatment for Sarcomas and Melanomas)
Brief Title: Using QPOP to Predict Treatment for Sarcomas and Melanomas
Status: Recruiting | Type: Observational
Sponsor: National Cancer Centre, Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: Q-SAM
Record Dates: First submitted 2021-07-27; First posted 2021-08-03 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Sarcoma; Melanoma
Keywords: Tumour-derived models; Organoids; Ex vivo drug testing; Personalised therapy; QPOP
MeSH Terms: conditions — Sarcoma; Melanoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumour Samples - Baseline upon study enrolment and on disease progression where clinically applicable.
  Enrolled patients undergoing a procedure where tumour tissue is removed for diagnostic or other clinical purposes, will be asked to donate any tissue that is in excess and not needed for diagnostic purposes, for this research study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a multi-cohort proof of concept study involving patients with sarcomas or melanomas. Patient models, both two- and three-dimensional, will be derived from tumour samples. These will then be used to evaluate drug sensitivities ex vivo.

Enrolled patients will undergo resections or biopsies as part of standard-of-care, which will be used to generate patient models. Patients will receive standard-of-care systemic treatment. Patient models will also be subjected up to a 14-drug screening panel. The majority of drugs in the respective drug panels has been shown to have activity in the respective cancers and would be used in the standard-of-care setting by treating physicians.

DETAILED DESCRIPTION:
Hypothesis: Ex vivo drug testing on patient-derived models using QPOP can identify drug sensitivities and combinations which may have clinical efficacy against sarcomas and melanomas.

Specific aim 1: To derive patient models, both two- and three-dimensional, of sarcomas and melanomas

Specific aim 2: To perform ex vivo drug testing on patient models of sarcoma and melanoma using QPOP

Specific aim 3: To assess the efficacy of phenotype directed therapy using QPOP to assign treatment after progression on standard-of-care treatment in sarcoma and melanoma

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of sarcoma or melanoma
* At least 1 tumour lesion amenable to fresh biopsy or resection
* Signed informed consent from patient or legal representative
* Able to comply with study-related procedures

Exclusion Criteria:

* There are no specific exclusion criteria if patients meet the inclusion criteria

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient aged between 21 to 99 diagnosed with sarcoma or melanoma.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-09-08 (Actual); Primary Completion 2028-10-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with successful model generation for each tumour subtype. | 8 years.
  Patients enrolled on study will undergo resection or biopsy of fresh tumour tissue to obtain cells for the generation of models.
Rates of radiological response from QPOP-directed treatment regimens. | 8 years.
  Complete and partial clinical response and stable disease.
Survival outcomes from QPOP-directed treatment regimens. | 8 years.
  Overall survival, progression-free survival.

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Shiwen Yang, BSc, MB BChir, PhD, Principal Investigator — National Cancer Centre, Singapore
Locations (1):
- National Cancer Centre Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No